CLINICAL TRIAL: NCT00496210
Title: Understanding Caregiver Adaptation to Pervasive Developmental Disorders
Brief Title: Predictors of Caregiver Adaptation to Pervasive Developmental Disorders
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907178; 07-HG-N178
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2015-12-07

CONDITIONS: Autism; Asperger's Syndrome; Rett's Disorder
Keywords: Adaptation; Pervasive Developmental Disorder; Autism Spectrum Disorders; Pervasive Developmental Disorders; Caregiver Adaptation
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Rett Syndrome; Child Development Disorders, Pervasive; Autism Spectrum Disorder

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will explore predictors of how caregivers might adapt to children diagnosed with a pervasive developmental disorder (PDD), including autism, Asperger s syndrome, childhood disintegrative disorder, Rett s disorder or other not specified PDD. PDD presents particular challenges for caregivers because of the communication and socialization challenges of affected children and because of the uncertainty surrounding the cause, prognosis and recurrence risks.

People 18 years of age or older who are the primary caregiver for a child diagnosed with a PDD may be eligible for this study. Participants fill out a survey, either online or in hard copy, that includes information in the following categories:

* How being a caregiver for a child with a PDD has impacted the caregiver.
* How much control the caregiver feels that he or she or others have over certain aspects of their child s PDD.
* What the caregiver thinks caused the child s PDD.
* What coping techniques the caregiver uses in caring for a child with a PDD.
* How uncertain the caregiver feels about his or her child s PDD.
* What the caregiver feels about him- or herself as a caregiver of a child with a PDD.
* General questions about the caregiver, his or her family and the child with a PDD.

DETAILED DESCRIPTION:
This study aims to understand the predictors of adaptation among primary caregivers of children with a pervasive developmental disorder (PDD). PDD presents particular challenges for caregivers because of the communication and socialization challenges of affected children, as well as the uncertainty surrounding the cause, prognosis and recurrence risks. The literature suggests that these challenges may make the process of adapting to having a child with a PDD different than it is for other chronic conditions. This study of caregivers is based on Lazarus and Folkman s Transactional Model of Stress and Coping. A cross-sectional design will be used to investigate the relationships among causal attributions, control perceptions, coping and adaptation. Caregivers will be recruited from support groups, listservs and magazines targeted to autism and other PDDs. Participants will be asked to complete either a web-based or paper survey. The main outcome measure is psychological adaptation to caregiving a child with PDD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Must be 18 or older and the primary caregiver for a child with one of the five diagnosis categorized as a pervasive developmental disorder.

EXCLUSION CRITERIA:

May not be younger than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2007-06-27; Study Completion 2015-12-07

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Affleck G, Tennen H, Pfeiffer C, Fifield J. Appraisals of control and predictability in adapting to a chronic disease. J Pers Soc Psychol. 1987 Aug;53(2):273-9. doi: 10.1037//0022-3514.53.2.273. PMID 3625467
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Aldwin CM, Revenson TA. Does coping help? A reexamination of the relation between coping and mental health. J Pers Soc Psychol. 1987 Aug;53(2):337-48. doi: 10.1037//0022-3514.53.2.337. PMID 3625471